CLINICAL TRIAL: NCT04627831
Title: Randomized Parallel Group Study Comparing the Renal Safety of CAPTISOL-Enabled™ Iohexol (CE-Iohexol) Injection and Omnipaque™ (Iohexol) Injection in Patients With Impaired Renal Function Undergoing Coronary Angiography
Brief Title: Comparison of Captisol-Enabled™ Iohexol and Omnipaque™ in Patients With Impaired Renal Function Undergoing Coronary Angiography
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal decision
Sponsor: Ligand Pharmaceuticals (Industry)
Collaborators: CyDex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CE-Iohexol - Study 201; Ligand 201 (Other: Ligand Pharmaceuticals); CAP201 (Other: Ligand Pharmaceuticals)
Record Dates: First submitted 2020-10-27; First posted 2020-11-13 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2021-02

CONDITIONS: Contrast-induced Nephropathy
MeSH Terms: interventions — Iohexol

STUDY DESIGN:
Intervention Model Description: Patients with impaired renal function scheduled for coronary angiography will be assessed for study eligibility. Prior to the planned coronary angiography procedure on Day 1, eligible patients will be randomized 1:1 to receive either CE-Iohexol Injection or iohexol. Randomization will be stratified by the following 2 factors.
  * Diabetes mellitus status:
    * Diabetics; or
    * Non-diabetics; and
  * Baseline eGFR, defined as the eGFR obtained as part of eligibility screening:
    * <45 mL/min/1.73 m2; or
    * 45 mL/min/1.73 m2.
  Contrast volumes will be determined according to medical need. All subjects will be well hydrated before and after the examination, according to good clinical practice and institution's standard procedures.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, and site personnel evaluating the subjects, will be blinded to the contrast media administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CE-Iohexol (Experimental): Subject is randomized to receive CE-Iohexol Injection
  Interventions: Drug: CE-Iohexol
- Omnipaque™ (Iohexol) (Active Comparator): Subject is randomized to receive Omnipaque™ Iohexol Injection
  Interventions: Drug: Iohexol

INTERVENTIONS:
Drug: CE-Iohexol — Captisol-Enabled™ Iohexol as needed for the diagnostic procedure. Volume will be determined according to medical need.
  Other Names: Captisol-Enabled™ Iohexol
  Arms: CE-Iohexol
Drug: Iohexol — Iohexol as needed for the diagnostic procedure. Volume will be determined according to medical need.
  Other Names: Omnipaque™ (Iohexol)
  Arms: Omnipaque™ (Iohexol)

SUMMARY:
Randomized parallel group study comparing the renal safety of Captisol-Enabled™ Iohexol (CE-Iohexol) Injection and Omnipaque™ (Iohexol) Injection in patients with impaired renal function undergoing coronary angiography.

DETAILED DESCRIPTION:
The purpose of this trial is to demonstrate a reduction in the incidence of contrast-induced acute kidney injury (CI-AKI), also known as contrast-induced nephropathy (CIN), and the equivalence of image quality following administration of Captisol-Enabled™-Iohexol (CE-Iohexol) Injection compared to Omnipaque™(Iohexol) Injection in patients with impaired renal function undergoing invasive coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years
2. Referred for a coronary angiography (with or without percutaneous coronary intervention) and must meet either 1 of the following criteria:

   1. Estimated glomerular filtration rate (eGFR) <45 and ≥15 mL/min/1.73 m2 as determined by the Chronic Kidney Disease Epidemiology Collaboration (CKD- EPI) equation; or
   2. eGFR <60 and ≥45 mL/min/1.73 m2 as determined by the CKD-EPI equation and at least 1 of the following conditions:

      * Age >75 years
      * Diabetes mellitus with glycosylated hemoglobin (HbA1c) ≤10%
      * New York Heart Association (NYHA) class II or III heart failure
      * Albuminuria with urine albumin-to-creatinine ratio (UACR) or urine protein-to- creatinine ratio (UPCR) ≥300 and ≤4000 mg/g; or
      * Anemia, with hemoglobin levels ≥8 g/dL but <12.0 g/dL in women and <13.0 g/dL in men, as defined by the World Health Organization
3. If female, must also meet any 1 of the following criteria:

   1. Surgically sterile with bilateral tubal ligation, bilateral salpingectomy, bilateral oophorectomy, or hysterectomy
   2. Postmenopausal with amenorrhea for at least 1 year and follicle-stimulating hormone in the postmenopausal range; or
   3. Is a woman of childbearing potential, non-pregnant and non-lactating at Screening, and must agree to use a protocol-recommended method of birth control or abstain from heterosexual intercourse, beginning at least 30 days prior to and until 30 days following investigational contrast agent administration
4. If a male who can father a child, must also meet all of the following criteria:

   1. Willing to use a protocol-recommended method of birth control, ie, a double barrier approach (eg, condoms with spermicide) or abstain from heterosexual intercourse with women of childbearing potential, from Day 1 until at least 90 days after investigational contrast agent administration; and
   2. Willing to refrain from sperm donation from Day 1 until at least 90 days after investigational contrast agent administration
5. Willing to undergo protocol-recommended blood and urine collections, physical examinations, and laboratory investigations; and
6. Willing and able to provide written informed consent

Exclusion criteria

1. eGFR <15 mL/min/1.73 m2
2. Reduction in eGFR by approximately 25% that is considered to be acute per the Investigator's judgment
3. Body weight >125 kg
4. Uncorrected clinically significant abnormalities of clinical laboratory assessments which, in the Investigator's opinion, will interfere with the study conduct, including but not limited to the following:

   1. HbA1c >10%
   2. Blood glucose >270 mg/dL
   3. Hemoglobin <8 g/dL
   4. Albuminuria with UACR or UPCR >4000 mg/g; or
   5. Aspartate aminotransferase or alanine aminotransferase >3 x upper limit of reference range
5. Positive test for severe acute respiratory syndrome coronavirus 2 RNA at Screening;
6. Positive test for human immunodeficiency virus antibody, hepatitis B surface antigen, or hepatitis C virus RNA at Screening
7. Uncontrolled hypertension, with systolic blood pressure (BP) >180 mmHg or diastolic BP >110 mmHg at Screening, based on the average of 3 BP measurements obtained from the patient's dominant arm
8. Hypotension, that is considered to be of recent occurrence per the Investigator's judgment, and required resuscitation with intravenous fluids
9. Non-cardiac acute illness or injuries that, in the opinion of the Investigator, could put the patient at risk or obscure the interpretation of the results of the study
10. Known allergy or sensitivity to iodinated contrast agents, Captisol, or any of the excipients in the study contrast agent that cannot be adequately managed with prophylactic treatment per the Investigator's judgment and Good Clinical Practice
11. Known allergy to heparin, history of heparin-induced thrombocytopenia, or history of heparin induced thrombocytopenia with thrombosis
12. Chronic disease(s) that, in the opinion of the Investigator, could interfere with (or for which the treatment might interfere with) the conduct of the study or interpretation of the study results or would place the patient at undue risk by participating in the study, including but not limited to the following:

    1. NYHA class IV or decompensated heart failure; or
    2. Cirrhosis of the liver
13. Inability to receive periprocedural intravenous volume expansion
14. Received contrast media within 10 days prior to the scheduled coronary angiography
15. Unable or not willing to come off non-steroidal anti-inflammatory drugs, including ibuprofen, for at least 24 hours before the scheduled procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of contrast-induced acute kidney injury (CI-AKI) | 7 days
  Evaluate the incidence of CI-AKI in patients with impaired renal function undergoing coronary angiography, from baseline to any blood draw within 7 days following intravascular administration of CE-iohexol compared with Omnipaque (iohexol).

SECONDARY OUTCOMES:
Image quality | Day 1
  Compare image quality of coronary angiography in patients administered CE-iohexol versus iohexol.
Change in serum creatinine (SCr) | 7 days
  Evaluate the changes in SCr in patients administered CE-iohexol versus iohexol.
Proportion of patients exhibiting an increase in SCr | 7 days
  Evaluate the proportion of patients exhibiting an increase in SCr following intravascular administration of CE-iohexol compared with iohexol.
Change in serum cystatin C | 7 days
  Evaluate the changes in serum cystatin C in patients administered CE-iohexol versus iohexol.
Incidence of Adverse Events | 30 days
  The number of patients with adverse events (AE) and serious adverse events will be assessed and graded according to Common Terminology Criteria for Adverse Events (CTCAE) v 4.0. Monitoring for Major Adverse Cardiac and Renal Events (MARCEs) will be part of the AE assessment.

OTHER OUTCOMES:
Change in novel biomarkers of renal injury | 7 days
  Evaluate the change in blood and urine biomarkers of renal injury from baseline to peak at 48 hours in patients administered CE-iohexol versus iohexol. Biomarkers may include neutrophil gelatinase-associated lipocalin, liver-type fatty acid binding protein and kidney injury molecule-1.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Marschke, PhD, Study Director — Ligand Pharmaceuticals